CLINICAL TRIAL: NCT01114997
Title: Effect of Lidocaine and Esmolol Alone or in Combination to Improve the Quality of Recovery, Maintaining Hemodynamic Stability During Abdominal Surgery
Brief Title: Effect of Lidocaine and Esmolol to Improve the Quality of Recovery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The early report didn't show any benefit.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Residency program director, Department of anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00020608
Record Dates: First submitted 2010-04-23; First posted 2010-05-03 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Pain; Constipation; Nausea; Vomiting
Keywords: Lidocaine Infusion; Esmolol Infusion; Anesthetic adjuvant; Abdominal surgery; Pain management; Hemodynamic stability; Perioperative outcomes
MeSH Terms: conditions — Pain; Constipation; Nausea; Vomiting; Agnosia | interventions — Lidocaine; esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lidocaine (Active Comparator): Pre-Induction: Lidocaine Loading: 1 mg/kg Post- Induction:Lidocaine Infusion: 12.5-25 mcg/kg/min 0.75-1.5 mg/kg/h)
  Interventions: Drug: Lidocaine
- Esmolol (Active Comparator): Pre-Induction: Loading dose 750 mcg/Kg (0.75 mg/kg) Post-Induction: Infusion dose 7.5 - 15 mcg /kg/min
  Interventions: Drug: Esmolol
- Lidocaine + Esmolol (Combo) (Experimental): Performed with the administration of both drugs.
  Pre-induction:
  Lidocaine Loading dose(1 mg/kg)+Esmolol Loading dose(750 mcg/Kg)
  Post-induction:
  Infusion rate: Lidocaine(12.5-25 mcg/kg/min) + Esmolol(7.5-15 mcg/kg/min)
  Interventions: Drug: Lidocaine + Esmolol (Combo)

INTERVENTIONS:
Drug: Lidocaine — Pre-Induction: Lidocaine Loading: 1 mg/kg After Induction:Lidocaine Infusion: 12.5-25 mcg/kg/min 0.75-1.5 mg/kg/h)
  Arms: Lidocaine
Drug: Esmolol — Esmolol Pre-Induction: Loading dose 750 mcg/Kg (0.75 mg/kg) Esmolol Post Induction: Infusion dose 7.5 - 15 mcg /kg/min
  Arms: Esmolol
Drug: Lidocaine + Esmolol (Combo) — Pre-induction: Lidocaine Loading dose(1 mg/kg) + Esmolol Loading dose(750 mcg/Kg)
  Maintenance Infusion rate after Induction:
  Lidocaine(12.5-25 mcg/kg/min) + Esmolol(7.5-15 mcg/kg/min)
  Arms: Lidocaine + Esmolol (Combo)

SUMMARY:
The purpose of this prospective, randomized, double-blinded, active-controlled study is:

To assess the effectiveness of systemic administration of lidocaine and esmolol in combination (vs. either drug alone) will result in improved postoperative outcomes for patients undergoing abdominal surgery (e.g., less pain and postoperative constipation, nausea and vomiting, faster return of bowel function, resumption of normal activities of daily living), leading to a shorten length of hospital stay, maintaining hemodynamic stability during general anesthesia, when administered as intravenous adjuvants

DETAILED DESCRIPTION:
Finding the optimal combination of anesthetic adjuvant drugs for maintaining hemodynamic stability during surgery is a challenge (1-3). Traditionally, potent opioid analgesics like fentanyl and its newer analogs have been used for this purpose. However, use of opioid compounds is associated with well-known side effects (e.g., ventilatory depression, postoperative nausea and vomiting, constipation, ileus, bladder dysfunction, urinary retention, pruritus, drowsiness and sedation). All of these common side effects interfere with the early recovery process and contribute to a delayed resumption of normal activities (4, 5). Increasingly, non-opioid analgesics (e.g. β-blockers and local anesthetics) are being utilized as adjuvant drugs during surgery for treatment of acute hyperdynamic responses (increased catecholamine release) during surgery, as well as, facilitation of the recovery process after surgery because of their anesthetic and analgesic-sparing effects. The β-blocking drugs, esmolol and labetalol have been used as an alternative to short-acting opioid analgesics for controlling the transient, acute autonomic responses during surgery (5-8), They have been shown to reduce the anesthetic requirement during intravenous (propofol) or volatile-based anesthesia (6,7,10-13) and to decrease opioid consumption intraoperatively and in the PACU (8). They may also improve hemodynamic stability during induction and emergence from anesthesia in the perioperative and early postoperative period and facilitate the resumption of normal activities after major surgical procedures. The anesthetic and analgesic-sparing effects of β -blockers also lead to a faster emergence from anesthesia and reduce postoperative opioid side effects (e.g., PONV) (14-18). Perioperative intravenous esmolol has shown improvement in perioperative outcomes, decreases acute hemodynamic responses, reduces anesthetics and opioids use during anesthesia, facilitates a faster emergence from anesthesia, reduces intraoperative and postoperative opioid requirements, reduces side effects as such as pruritus, constipation, ileus, nausea and vomiting (PONV) and thereby shortens the hospital stay. (3, 7, 13, 18)

Local anesthetics like lidocaine possess analgesic, antihyperalgesic and anti-inflammatory properties. Perioperative intravenous lidocaine has shown improvement in perioperative outcomes in patients undergoing abdominal surgery to decrease intraoperative requirement of Inhalants/Intravenous agents, opioid consumption, postoperative pain, fatigue, nausea and vomiting scores, maintain hemodynamic stability, facilitate a more rapid recovery of gastrointestinal function, improve postoperative recovery, fast resumption of normal activities of daily living and shorten length of hospital stay, when administered as an adjuvant during surgery.(19,23-29,33)

Theoretically, it would be extremely beneficial to administer an adjuvant (to patients undergoing abdominal surgery) that is capable of effectively controlling autonomic responses during surgery, while providing a faster recovery with fewer side effects. Preliminary data suggests that the perioperative effects of systemic administration of lidocaine and esmolol is most effective in facilitating bowel recovery, decreasing opioid consumption in the intra/postoperative period, and shorten length of hospital stay with early recovery. Therefore, we designed this prospective, randomized, double-blinded, active-controlled study to test the hypothesis that systemic administration of lidocaine and esmolol in combination (vs. either drug alone) for maintenance of hemodynamic stability during surgery will result in improved postoperative outcomes for patients undergoing abdominal surgery (e.g., less pain and postoperative nausea and vomiting, and faster return of bowel function and resumption of normal activities of daily living); leading to a shorten length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo abdominal surgical procedures
* Willingness and ability to sign an informed consent document
* No allergies to anesthetic or analgesic medications
* 18 - 80 years of age
* American Society of Anesthesiologists (ASA) physical status classification: Class I - III adults of either sex
* Women of childbearing potential must be currently practicing an acceptable form of birth control, and have a negative urine or blood pregnancy test
* Patients with systolic blood pressure greater than 80 and less than 150 at baseline, diastolic blood pressure less than 100 at baseline.

Exclusion Criteria:

* Inability to comprehend the pain assessment tools.
* Patients with known allergy, hypersensitivity or contraindications to anesthetic or analgesic medications
* Patients with clinically-significant medical conditions, such as brain, heart, kidney, endocrine, or liver diseases,
* Peptic ulcer disease or bleeding disorders
* Patients with history of hepatic, renal, cardiac failure, organ transplant, or diabetes
* Patients with reactive airway disease (asthma)
* Patients with seizures
* Chronic use of ß-blocker or calcium channel blocker
* Morbid obesity (body mass index >40)
* Pregnant or lactating women
* Subjects with a history of alcohol or drug abuse within the past 3 months
* Any other conditions or use of any medication which may interfere with the conduct of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Esmolol: Pre-Induction:
  Esmolol Loading dose: 750 mcg/Kg (0.75 mg/kg)
  Post-Induction:
  Infusion dose 7.5 - 15 mcg /kg/min
- Lidocaine + Esmolol (Combo): Pre-induction:
  Lidocaine Loading dose(1 mg/kg)+Esmolol Loading dose(750 mcg/Kg)
  Post-induction:
  Infusion rate: Lidocaine(12.5-25 mcg/kg/min) + Esmolol(7.5-15 mcg/kg/min)
Period: Overall Study
Arm/Group | Lidocaine | Esmolol | Lidocaine + Esmolol (Combo)
Started | 11 | 10 | 11
Completed | 11 | 10 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lidocaine: Pre-Induction:
  Lidocaine Loading: 1 mg/kg
  Post- Induction:
  Lidocaine Infusion: 12.5-25 mcg/kg/min 0.75-1.5 mg/kg/h)
- Lidocaine + Esmolol (Combo): Pre-induction:
  Lidocaine Loading dose(1 mg/kg)+Esmolol Loading dose(750 mcg/Kg)
  Post-Induction (Maintenance Infusion):
  Lidocaine(12.5-25 mcg/kg/min) + Esmolol(7.5-15 mcg/kg/min)
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Esmolol | Lidocaine + Esmolol (Combo) | Total
Number analyzed (Participants) | 11 | 10 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (8) | 44 (3) | 38 (10) | 41 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 11 | 32
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — California, United States
  participants
    United States | 11 | 10 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Pain
Description: Outcome had a duration of one day at post-anesthesia care unit (PACU) Postoperative pain measured using a Verbal Rating Scale (VRS) Postoperative pain VRS scores: 0 = none pain to 10 = intolerable pain.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Lidocaine | Esmolol | Lidocaine + Esmolol (Combo)
Number analyzed (Participants) | 11 | 10 | 11
Score on a scale | 4 (4) | 2 (2) | 4 (3)

2. Primary Outcome: Number of Participants With Post Operative Pain One Month After Surgery
Description: Highest Post Operative pain one month after surgery, using a verbal rating score from 0 (no pain) to 10 (highest level of pain).
  Patient received a post-operative follow-up call one month after surgery.
Time Frame: 1 month
Population: Experience of pain at home
Measure: Number; unit: participants
Arm/Group | Lidocaine | Esmolol | Lidocaine + Esmolol (Combo)
Number analyzed (Participants) | 11 | 10 | 11
participants | 10 | 8 | 10

3. Secondary Outcome: Opioid Consumption Obtained From the Recorded Data
Description: Postoperative use of opioid consumption inside hospital (recorded by study staff and data obtained from patient charts)
Time Frame: 1 day
Population: Opioid: Hydromorphone
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Lidocaine | Esmolol | Lidocaine + Esmolol (Combo)
Number analyzed (Participants) | 11 | 10 | 11
mg | 1.5 (1) | 1 (0.8) | 1.5 (1)

4. Secondary Outcome: Number of Participants With Postoperative Nausea One Day After Surgery
Description: Postoperative nausea using a Verbal Rating Scale Outcomes measured at the first day after surgery
Time Frame: 1day
Measure: Number; unit: participants
Arm/Group | Lidocaine | Esmolol | Lidocaine + Esmolol (Combo)
Number analyzed (Participants) | 11 | 10 | 11
participants | 3 | 2 | 3

5. Secondary Outcome: Return to Normal Activities of Daily Living Using Follow up Questionnaires
Description: Description: return to normal activities of daily living(including dietary intake, bowel and bladder function, physical activities)
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Lidocaine | Esmolol | Lidocaine + Esmolol (Combo)
Number analyzed (Participants) | 11 | 10 | 11
participants | 10 | 8 | 8

6. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction using a verbal rating scale from 0 to 10 0= Not satisfied 10= Excellent
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Lidocaine + Esmolol (Combo): Pre-induction:
  Lidocaine Loading dose(1 mg/kg)+Esmolol Loading dose(750 mcg/Kg)
  Post-induction:
  Infusion rate: Lidocaine (12.5-25 mcg/kg/min) + Esmolol (7.5-15 mcg/kg/min)
Arm/Group | Lidocaine | Esmolol | Lidocaine + Esmolol (Combo)
Number analyzed (Participants) | 11 | 10 | 11
Score on a scale | 9.4 (0.8) | 9.2 (1) | 8.3 (2)

7. Secondary Outcome: Post-anesthesia Care Unit (PACU) Stay
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Lidocaine | Esmolol | Lidocaine + Esmolol (Combo)
Number analyzed (Participants) | 11 | 10 | 11
Minutes | 236 (147) | 116 (38) | 214 (125)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Lidocaine | Esmolol | Lidocaine + Esmolol (Combo)
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No